CLINICAL TRIAL: NCT06020937
Title: Olfactory and Trigeminal Functions in Patients With Multiple Sclerosis
Brief Title: Olfactory and Trigeminal Functions in Patients With Multiple Sclerosis: Case-control Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Catania (Other)
Collaborators: University of Roma La Sapienza (Other); Hospital General Universitario Santa Lucia (Other); Klinik und Poliklinik fur Kinderheilkunde (Other)
Responsible Party: Principal Investigator, Arianna Di Stadio, Associate Professor (temporary), University of Catania
Other Study IDs: UniCT192023
Record Dates: First submitted 2023-08-22; First posted 2023-09-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Healthy patients
  Interventions: Diagnostic Test: TDI; Diagnostic Test: Trigeminal Test; Diagnostic Test: Visual Analogue Scale Ratings; Diagnostic Test: Quality of smell Questionnaire
- Multiple Sclerosis 1: Patients with multiple Sclerosis and Trigeminal disorders
  Interventions: Diagnostic Test: TDI; Diagnostic Test: Trigeminal Test; Diagnostic Test: Cognitive Evaluation by Montreal Cognitive Assessment; Diagnostic Test: Anxiety and Depression questionnaire; Diagnostic Test: Visual Analogue Scale Ratings; Diagnostic Test: Quality of smell Questionnaire
- Multiple Sclerosis 2: Patients with Multiple Sclerosis without trigeminal concerns
  Interventions: Diagnostic Test: TDI; Diagnostic Test: Trigeminal Test; Diagnostic Test: Cognitive Evaluation by Montreal Cognitive Assessment; Diagnostic Test: Anxiety and Depression questionnaire; Diagnostic Test: Visual Analogue Scale Ratings; Diagnostic Test: Quality of smell Questionnaire

INTERVENTIONS:
Diagnostic Test: TDI — Sniffin' Sticks Threshold and Identification Test
Diagnostic Test: Trigeminal Test — Test the trigeminal smell answer by a device that releases air and a substance that stimulates the trigeminal response
Diagnostic Test: Cognitive Evaluation by Montreal Cognitive Assessment — Montreal Cognitive assessment
  Groups: Multiple Sclerosis 1; Multiple Sclerosis 2
Diagnostic Test: Anxiety and Depression questionnaire — Specific test to evaluate patient's mood
  Groups: Multiple Sclerosis 1; Multiple Sclerosis 2
Diagnostic Test: Visual Analogue Scale Ratings — * Smell ability (How is your sense of smell right now? 0 cannot smell, 1-3 severe impairment, 4-6 moderate impairment, 7-9 mild impairment, 10 normal)
  * Nasal breathing (How well can you breathe through your nose right now? 0 complete nasal obstruction, 1-3 severe impairment, 4-6 moderate impairment, 7-9 mild impairment, 10 normal)
Diagnostic Test: Quality of smell Questionnaire — Patients will answer to a validated questionnaire

SUMMARY:
The sensation of smell is influenced by the somatosensory and chemesthetic sensati¬ons of the nose: for example, the cooling sensation of menthol or the prickle of carbon dioxide from carbonated drinks. These sensations are mediated in the nose by the trigeminal nerve and there is increasing evidence that trigeminal and olfactory functions are closely linked and potentially interdependent. In addition, trigeminal activation is crucial to the perception of nasal airflow. Some researchers speculate about the impact of trigeminal nerve on the entire olfactory sensation and about the presence of some specific "trigeminal cells" into the nose.Patients with Multiple sclerosis (MS) can suffer from quantitative olfactory disorders that generally are of light entity and do not interfere with daily life activities but it is important to underline that olfactory loss can be an onset sign of the MS. Considering the "trigeminal component" in the olfaction, because trigeminal nerve inflammation is quite common in MS patients due to central and peripheral inflammation, it could be possible that these patients suffer from changes in the quantitative, but more in the qualitative smell functions that are generally not identified because poorly investigated.

DETAILED DESCRIPTION:
From a theoretically point of view pain in the trigeminal nerve increases the surrounding perception, including the perception of the odors. It has been shown that by using sweet food it is possible to reduce the level of pain; on the other side, sweet food in contrast to the bitter one was able to reduce the sensation of odor unpleasantness present with pain increase.

To date no studies have investigated the relationship between trigeminal inflammation, odors and pain in a cohort of patients with MS. This study aims at investigating the possible correlation between alteration in trigeminal functions and perception of odors using Sniffin' Stick Threshold, Detection and Identification test and quality smell questionnaire in a sample of healthy patients compared to MS patients.

ELIGIBILITY:
Inclusion Criteria:

Adult women (age 18 to 55) diagnosed with multiple sclerosis using the 2017 McDonald Criteria under treatment with Disease Modifying Therapy (DMTs) with or without trigeminal concerns, or newly diagnosed with MS

Exclusion Criteria:

* Chronic rhinosinusitis with and without nasal polyposis; current allergic rhinitis; other nasal issues that lead to olfactory dysfunction
* anamnestic COVID with incomplete recovery
* Neurodegenerative disorders (Parkinson, Alzheimer, Fronto-temporal Dementia, cognitive impairment and brain vascular diseases)
* History of stroke in the last three years
* Depression or any psychiatric condition
* intake of drugs with sedating side effects
* major health issues that might affect olfactory function (e.g., significant renal insufficiency, uncontrolled diabetes)
* Chronic alcoholism / drug abuse
* Severe head trauma
* Severe facial injuries
* Smoker over 20 cigarettes day or smoking from more than 15 years

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Number of participants: 400, 200 healthy controls, and 200 patients diagnosed with multiple sclerosis divided as follow: 100 with manifest trigeminal pain 100 without known trigeminal pathology.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Trigeminal component | 12 months
  One bottle contains 10ml Eucalyptol (pure / 99%), the other bottle contains only air 15ml stimuli would be released from both bottles using the squeezer device A 3cm long, 4mm inner diameter silicon tubing is placed over the nozzle of each bottle to minimize irritation at the nostrils Silicon tubing should reach beyond the nasal valve area
  * Trigeminal intensity ratings (How intense is the tickling or cool sensation in the nose? 0 no feeling, 10 very strong feeling)
  * The trial can be done on the left nostril, then on the right nostril and this already corresponds to the first presentation for the actual test
    * Total of 20 presentations (10 on each side) with interstimulus interval of around 10 seconds between each presentation, and a longer pause of 30 seconds every 5 presentations
    * The score is the sum of correct lateralizations

CONTACTS AND LOCATIONS:
Locations (1):
- Arianna Di Stadio, Catania, Sicily, Italy

IPD SHARING:
Plan to Share IPD: Undecided
History collection
  Magnetic Resonance Imaging (MRI) 1.5-T Signal scanner; Whole brain scan; T2 FLAIR and double-echo long-TR axial, 3-mm axial and 1mm coronal slices; Olfactory bulb volumetrics
  "Sniffin' Sticks" Threshold and Identification Test Perform monorhinal
  Visual Analogue Scale Ratings Smell ability (How is your sense of smell right now? 0 cannot smell, 1-3 severe impairment, 4-6 moderate impairment, 7-9 mild impairment, 10 normal) Nasal breathing (How well can you breathe through your nose right now? 0 complete nasal obstruction, 1-3 severe impairment, 4-6 moderate impairment, 7-9 mild impairment, 10 normal)
  Quality of smell Questionnaire
  Cognitive Evaluation by Montreal Cognitive Assessment
  Anxiety and Depression questionnaire
  Trigeminal Lateralization

REFERENCES:
- [Background] Hummel T, Frasnelli J. The intranasal trigeminal system. Handb Clin Neurol. 2019;164:119-134. doi: 10.1016/B978-0-444-63855-7.00008-3. PMID 31604542
- [Background] Frasnelli J, Manescu S. The intranasal trigeminal system. In: Buettner A, editor. Dordrecht; 2017. p. 881-95
- [Background] Hummel T, Iannilli E, Frasnelli J, Boyle J, Gerber J. Central processing of trigeminal activation in humans. Ann N Y Acad Sci. 2009 Jul;1170:190-5. doi: 10.1111/j.1749-6632.2009.03910.x. PMID 19686136
- [Background] Daiber P, Genovese F, Schriever VA, Hummel T, Mohrlen F, Frings S. Neuropeptide receptors provide a signalling pathway for trigeminal modulation of olfactory transduction. Eur J Neurosci. 2013 Feb;37(4):572-82. doi: 10.1111/ejn.12066. Epub 2012 Dec 3. PMID 23205840
- [Background] Doty RL, Brugger WE, Jurs PC, Orndorff MA, Snyder PJ, Lowry LD. Intranasal trigeminal stimulation from odorous volatiles: psychometric responses from anosmic and normal humans. Physiol Behav. 1978 Feb;20(2):175-85. doi: 10.1016/0031-9384(78)90070-7. No abstract available. PMID 662939
- [Background] Mihara S, Shibamoto T. The role of flavor and fragrance chemicals in TRPA1 (transient receptor potential cation channel, member A1) activity associated with allergies. Allergy Asthma Clin Immunol. 2015 Mar 16;11(1):11. doi: 10.1186/s13223-015-0074-0. eCollection 2015. PMID 25897313
- [Background] Scheibe M, Schulze S, Mueller CA, Schuster B, Hummel T. Intranasal trigeminal sensitivity: measurements before and after nasal surgery. Eur Arch Otorhinolaryngol. 2014 Jan;271(1):87-92. doi: 10.1007/s00405-013-2466-4. Epub 2013 Apr 9. PMID 23568039
- [Background] Zhao K, Jiang J, Blacker K, Lyman B, Dalton P, Cowart BJ, Pribitkin EA. Regional peak mucosal cooling predicts the perception of nasal patency. Laryngoscope. 2014 Mar;124(3):589-95. doi: 10.1002/lary.24265. Epub 2013 Jun 28. PMID 23775640
- [Background] Li C, Farag AA, Maza G, McGhee S, Ciccone MA, Deshpande B, Pribitkin EA, Otto BA, Zhao K. Investigation of the abnormal nasal aerodynamics and trigeminal functions among empty nose syndrome patients. Int Forum Allergy Rhinol. 2018 Mar;8(3):444-452. doi: 10.1002/alr.22045. Epub 2017 Nov 22. PMID 29165896
- [Background] Konstantinidis I, Tsakiropoulou E, Chatziavramidis A, Ikonomidis C, Markou K. Intranasal trigeminal function in patients with empty nose syndrome. Laryngoscope. 2017 Jun;127(6):1263-1267. doi: 10.1002/lary.26491. Epub 2017 Feb 22. PMID 28224626
- [Background] Atalar AC, Erdal Y, Tekin B, Yildiz M, Akdogan O, Emre U. Olfactory dysfunction in multiple sclerosis. Mult Scler Relat Disord. 2018 Apr;21:92-96. doi: 10.1016/j.msard.2018.02.032. Epub 2018 Mar 3. PMID 29529530
- [Background] Zorzon M, Ukmar M, Bragadin LM, Zanier F, Antonello RM, Cazzato G, Zivadinov R. Olfactory dysfunction and extent of white matter abnormalities in multiple sclerosis: a clinical and MR study. Mult Scler. 2000 Dec;6(6):386-90. doi: 10.1177/135245850000600605. PMID 11212134
- [Background] da Silva CJ, da Rocha AJ, Mendes MF, Maia AC Jr, Braga FT, Tilbery CP. Trigeminal involvement in multiple sclerosis: magnetic resonance imaging findings with clinical correlation in a series of patients. Mult Scler. 2005 Jun;11(3):282-5. doi: 10.1191/1352458505ms1186oa. PMID 15957508
- [Background] Riello M, Cecchini MP, Zanini A, Di Chiappari M, Tinazzi M, Fiorio M. Perception of phasic pain is modulated by smell and taste. Eur J Pain. 2019 Nov;23(10):1790-1800. doi: 10.1002/ejp.1453. Epub 2019 Jul 29. PMID 31291496
- [Result] Di Stadio A, Bernitsas E, La Mantia I, Brenner MJ, Ralli M, Vaira LA, Colizza A, Cavaliere C, Laudani M, Frohman TC, De Vincentiis M, Frohman EM, Altieri M. Targeting Neuroinflammation to Alleviate Chronic Olfactory Dysfunction in Long COVID: A Role for Investigating Disease-Modifying Therapy (DMT)? Life (Basel). 2023 Jan 13;13(1):226. doi: 10.3390/life13010226. PMID 36676175